CLINICAL TRIAL: NCT01947608
Title: An Open-label, Multi-center, Expanded Treatment Protocol (ETP) of Oral LDK378 in Adult Patients With Non-small Cell Lung Cancer (NSCLC) Characterized by ALK Positivity
Brief Title: Expanded Treatment Protocol With LDK378 in ALK(+) NSCLC
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLDK378A2402
Record Dates: First submitted 2013-09-17; First posted 2013-09-20 (Estimated); Last update posted 2020-11-03 (Actual); Status verified 2019-12

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ceritinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: LDK378 — 750 mg. orally

SUMMARY:
Novartis-sponsored, open-label, multi-center, interventional ETP to provide LDK378 to patients with ALK (+)NSCLC, who have been pre-treated with an ALK inhibitor; except in countries where ALK inhibitors are not approved or available. The protocol will further evaluate the safety of LDK378 in patients with ALK(+) NSCLC.

ELIGIBILITY:
Inclusion Criteria (patients eligible for inclusion in this early treatment protocol have to meet all of the following criteria):

1. Histologically or cytologically confirmed diagnosis of NSCLC that demonstrates ALK positivity as assessed by approved FISH test (Abbott Molecular Inc), using Vysis breakapart probes (defined as 15% or more positive tumor cells); or the Ventana IHC test. If documentation of ALK positivity is not available, the test to confirm ALK positivity must be performed according to the above criterion, using a new tumor biopsy obtained prior to the first dose of ETP treatment (LDK378).
2. Stage IIIB or IV NSCLC patient with documented disease progression at enrollment, and who does not qualify or have access to LDK378 through a clinical trial.
3. Age 18 years or older at the time of informed consent.
4. WHO performance status 0-3.
5. Patients who have been pre-treated with an ALK inhibitor for locally advanced or metastatic NSCLC. Patients may be enrolled without prior exposure to an ALK inhibitor in countries where ALK inhibitors are not approved or available. Exposure to prior chemotherapy is not required.
6. Patients must have recovered from all toxicities related to prior anticancer therapies to grade ≤ 2 (CTCAE v 4.03), provided that concomitant medication is given prior to initiation of treatment with LDK378. Exception to this criterion: patients with any grade of alopecia are allowed to enter the treatment.
7. The following laboratory criteria have been met:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L
   * Hemoglobin (Hgb) ≥ 8 g/dL
   * Platelets ≥ 75 x 109/L
   * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN), except for patients with Gilbert's syndrome who may be included if total bilirubin ≤ 3.0 x ULN and direct bilirubin ≤ 1.5 x ULN
   * Aspartate transaminase (AST) < 3.0 x ULN, except for patients with liver metastasis, who are only included if AST < 5 x ULN; alanine transaminase (ALT) < 3.0 x ULN, except for patients with liver metastasis, who are only included if ALT < 5 x ULN.
   * Calculated or measured creatinine clearance (CrCL) ≥ 30 mL/min
8. Patient must have the following laboratory values or have the following laboratory values corrected with supplements to be within normal limits at screening:

   * Potassium ≥ LLN
   * Magnesium ≥ LLN
   * Phosphorus ≥ LLN
   * Total calcium (corrected for serum albumin) ≥ LLN
9. Written informed consent for the ETP protocol must be obtained prior to any screening procedures. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness.
10. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other ETP procedures.

Exclusion Criteria (patients eligible for this ETP must not meet any of the following criteria):

1. Patients with known hypersensitivity to any of the excipients of LDK378 (microcrystalline cellulose, mannitol, crospovidone, colloidal silicon dioxide and magnesium stearate).
2. Patients with symptomatic CNS metastases who are neurologically unstable or have required increasing doses of steroids within the 1 week prior to ETP entry to manage CNS symptoms.
3. Prior therapy with LDK378.
4. The patient is less than 5 half-lives from prior ALK inhibitor or targeted therapy (for adequate wash-out) without recovery from treatment toxicities to ≤ grade 1 or to their pretreatment levels.
5. Chemotherapy or an investigational therapy ≤ 3 weeks prior to starting the LDK378 treatment who have not recovered from side effects of such treatment toxicities to ≤ grade 2 or to their pre- treatment toxicities levels, with the exception of liver and cardiac functions which must be ≤ grade 1.
6. Patients who have received thoracic radiotherapy to lung fields ≤ 4 weeks prior to starting the study treatment or patients who have not recovered from radiotherapy-related toxicities. For all other anatomic sites (including radiotherapy to thoracic vertebrae and ribs) radiotherapy ≤ 2 weeks prior to starting the LDK378 treatment or have not recovered from radiotherapy-related toxicities. Palliative radiotherapy for bone lesions ≤ 2 weeks prior to starting LDK378 treatment is allowed.
7. Major surgery (e.g., intra-thoracic, intra-abdominal or intra-pelvic) within 4 weeks prior (2 weeks for resection of brain metastases) to starting LDK378 treatment or who have not recovered from side effects of such procedures. Video-assisted thoracic surgery (VATS) and mediastinoscopy will not be counted as major surgery, and patients can be enrolled in the ETP ≥ 2 weeks after the procedure.
8. Presence or history of a malignant disease other than NSCLC that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
9. Patients with known history of extensive disseminated bilateral interstitial fibrosis or interstitial lung disease, including a history of pneumonitis, hypersensitivity pneumonitis, interstitial pneumonia, obliterative bronchiolitis, and clinically significant radiation pneumonitis (i.e. affecting activities of daily living or requiring therapeutic intervention).
10. Patient has clinically significant, uncontrolled heart disease and/or recent cardiac event (within 6 months), such as:

    * unstable angina within 6 months prior to screening;
    * myocardial infarction within 6 months prior to screening;
    * history of documented congestive heart failure (New York Heart Association functional classification III-IV);
    * uncontrolled hypertension defined by a Systolic Blood Pressure (SBP) ≥ 160 mm Hg and/or Diastolic Blood Pressure (DBP) ≥ 100 mm Hg, with or without antihypertensive medication -
    * initiation or adjustment of antihypertensive medication(s) is allowed prior to screening;
    * ventricular arrhythmias; supraventricular and nodal arrhythmias not controlled with medication;
    * other cardiac arrhythmia not controlled with medication;
    * corrected QTc > 450 msec using Fridericia correction on the screening ECG
11. Impaired GI function or GI disease that may alter absorption of LDK378 or inability to swallow up to five LDK378 capsules daily
12. Ongoing GI adverse events > grade 2 (e.g. nausea, vomiting, or diarrhea) at the start of the ETP.
13. Receiving medications that meet one of the following criteria and that cannot be discontinued at least 1 week prior to the start of treatment with LDK378 and for the duration of the ETP participation (see Appendix 1: Tables 14-1, Table 14-2, Table 14-3, and Table 14-4):

    * Medication with a known risk of prolonging the QT interval or inducing Torsades de Pointes (please refer to http://www.azcert.org/medical-pros/drug-lists/drug-lists.cfm)
    * Strong inhibitors or strong inducers of CYP3A4/5 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
    * Medications with a low therapeutic index that are primarily metabolized by CYP3A4/5, CYP2C8 and/or CYP2C9 (please refer to http://medicine.iupui.edu/flockhart/table.htm or http://www.druginteractioninfo.org)
    * Therapeutic doses of warfarin sodium (Coumadin) or any other coumadin-derived anti-coagulant. Anticoagulants not derived from warfarin are allowed (eg, dabigatran, rivaroxaban, apixaban).
    * Unstable or increasing doses of corticosteroids
    * enzyme-inducing anticonvulsive agents
    * herbal supplements
14. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
15. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 3 months after the last dose of study treatment.

    In case of use of oral contraception, women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g., age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks prior to screening. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
16. Sexually active males unless they use a condom during intercourse while taking drug and for 3 months after the last dose of study treatment. Male patients for 3 months should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (46):
- United States (27):
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Banner MDACC, Gilbert, Arizona
  - Western Regional Medical Center, Inc., Goodyear, Arizona
  - Highlands Oncology Group, Fayetteville, Arkansas
  - City of Hope National Medical Center, Duarte, California
  - Moores UCSD Cancer Center, La Jolla, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Stanford University, Stanford, California
  - Eastern Connecticut Hematology & Oncology Associates, Norwich, Connecticut
  - Advanced Medical Specialties, Miami, Florida
  - Peachtree Hematology/Oncology Consultants, Atlanta, Georgia
  - Emory University School of Medicine/Winship Cancer Institute, Atlanta, Georgia
  - Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Indiana University Health Goshen Center for Cancer, Goshen, Indiana
  - Johns Hopkins Bayview Hospital, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Rockville, Maryland
  - Massachusetts General Hospital Mass General, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Jackson Oncology Associates, Jackson, Mississippi
  - Nebraska Cancer Specialist/Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mercy Clinic Oklahoma Communities Mercy Oncology, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - University of Utah / Huntsman Cancer Institute, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Argentina (3):
  - Novartis Investigative Site, CABA, Buenos Aires
  - Novartis Investigative Site, Buenos Aires, Buenos Aires F.D.
  - Novartis Investigative Site, Córdoba, Córdoba Province
- Colombia (2):
  - Novartis Investigative Site, Cali, Valle del Cauca Department
  - Novartis Investigative Site, Montería
- Hong Kong (2):
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Kowloon
- Novartis Investigative Site, Delhi, India
- Novartis Investigative Site, Amman, Jordan
- Mexico (2):
  - Novartis Investigative Site, Mexico City, Mexico City
  - Novartis Investigative Site, Mexico D F, Mexico City
- Philippines (2):
  - Novartis Investigative Site, City of Taguig, National Capital Region
  - Novartis Investigative Site, Quezon City
- South Korea (5):
  - Novartis Investigative Site, Bundang Gu, Gyeonggi-do
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Novartis Investigative Site, Bangkok, Thailand